CLINICAL TRIAL: NCT02618772
Title: Atomized Intranasal Midazolam for Anxiolysis and Facilitation of Laceration Repair in the Pediatric Emergency Department: A Randomized Controlled Trial
Brief Title: Intranasal Midazolam for Treatment of Anxiety in Children Undergoing Suturing in the Pediatric Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jennifer Turnbull, Dr. Jennifer Turnbull, MD, FRCPC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PED-08-053
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Anxiety; Lacerations
Keywords: Pediatrics; Laceration; Anxiety; Anti-Anxiety Agents
MeSH Terms: conditions — Anxiety Disorders; Lacerations | interventions — Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Saline (Placebo Comparator): 0.08ml/kg of saline to a maximum of 2ml intranasally with an atomizer MAD-300
  Interventions: Drug: Saline
- Intranasal Midazolam (Active Comparator): 0.08ml/kg (0.4mg/kg of 5mg/ml IV solution) intranasal midazolam, to a maximum of 2ml (10mg), with an atomizer MAD-300
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Intranasal administration of midazolam at dose of 0.4mg/kg (max 10 mg) one time 10 minutes prior to laceration repair
  Arms: Intranasal Midazolam
Drug: Saline — Intranasal administration of saline at a dose of 0.08ml/kg (max 2ml) one time prior to laceration repair as a placebo
  Arms: Intranasal Saline

SUMMARY:
Laceration repair can cause significant anxiety in children. As open wounds account for 21-25% of injuries in children presenting to the emergency department, the management of anxiety is of great importance. Anxiety can often lead to poor patient cooperation and the use of potentially excessive physical restraint. High rates of procedural anxiety have also been correlated with increased rates of negative behaviours after discharge.

The current standard of care for suture closure of lacerations throughout most of Canada is to provide local analgesia only. The literature has therefore focused on finding anxiolytic adjuncts to local analgesia.

Midazolam is an ideal adjunct due to its fast onset and short duration of action with an excellent safety profile. The advantages of the IN route are less pain on administration when compared to the IV and IM routes, and increased acceptability compared to the rectal route in older children. Oral midazolam also has poor palatability.

While the onset of INM at 5-10 minutes, and duration of 20-40 minutes make it an ideal candidate for anxiolysis in the ED its use has been limited by the common side effect of nasal irritation, burning and lacrimation when it is administered in its droplet form. The recent development of mucosal atomization devices (MAD) has resolved this issue by delivering 30-μ particles to the nasal mucosa.

Previous studies investigating the use of INM for laceration repair in the pediatric ED have demonstrated that INM is safe but most used non-validated measurement tools to assess anxiety and facilitation. Only one of these studies used atomized INM, retrospectively examining safety as the primary outcome. The authors reported an excellent safety profile for INM using the mucosal atomization device MAD-300 (Wolfe Tory Medical Inc.). The use of atomized INM for anxiolysis during pediatric laceration repair has not been evaluated prospectively.

Most studies have focused on preschool aged children (<6 years). While studies have demonstrated that the prevalence of procedural anxiety is higher in younger children, up to 51% of children age 7-12 years experience high levels of procedural distress. The effectiveness of INM in the pre-adolescent age group is, therefore, yet to be determined.

It is hypothesized that INM will reduce anxiety in children age 2-12 years undergoing laceration repair and will facilitate the successful completion of suturing by the physician.

ELIGIBILITY:
Inclusion Criteria:

* children 2-12 years requiring laceration repair using suturing and use of injected lidocaine

Exclusion Criteria:

* Administration in ER of analgesia or sedation other than acetaminophen or ibuprofen prior to enrolment
* ASA of III or greater
* Multi-system trauma
* Severe neurologic impairment or non-verbal autism, known allergy/hypersensitivity to lidocaine or midazolam
* Parent/guardian does not speak one of French or English
* No parent/guardian present during procedure

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2010-01; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on January 13, 2010 and was completed on March 17, 2015. Recruitment took place solely in the Pediatric Emergency Department at the Montreal Children's Hospital.
Groups:
- Intranasal Saline: 0.08ml/kg of saline to a maximum of 2ml intranasally with an atomizer MAD-300
  Saline: Intranasal administration of saline at a dose of 0.08ml/kg (max 2ml) one time prior to laceration repair as a placebo, 10 minutes prior to laceration repair
Period: Overall Study
Arm/Group | Intranasal Saline | Intranasal Midazolam
Started | 39 | 40
Withdrawal by Subject | 1 (The participant's family withdrew from the study after administration of the trial intervention.) | 0
Completed | 38 | 40
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study Population: Children 2-12 years old who presented to the Montreal Children's Hospital Emergency Department with a laceration requiring repair with sutures under local analgesia (local injection of lidocaine).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Saline | Intranasal Midazolam | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Customized [Mean (Standard Deviation); unit: years] — This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  years
    Intention to Treat (ITT): (n = 39, 40, 79) | 7.3554 (3.2152) | 6.8642 (3.5191) | 7.1067 (3.35997)
    Per-Protocol (PP): (n = 35, 37, 72) | 7.3848 (3.1826) | 6.8454 (3.6318) | 7.1076 (3.4077)
Sex/Gender, Customized [Number; unit: participants] — This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  participants
    Intention to Treat (ITT): Female | 10 | 15 | 25
    Intention to Treat (ITT): Male | 29 | 25 | 54
    Per-Protocol (PP): Female | 9 | 15 | 24
    Per-Protocol (PP): Male | 26 | 22 | 48
Region of Enrollment [Number; unit: Participants] — All participants were enrolled at the Montreal Children's Hospital in Montreal, Quebec (Canada). The address is as follows: 2300 Tupper, Montreal (QC), Canada, H3H 1P3.
  Participants
    Canada | 39 | 40 | 79
Laceration Length (cm) [Mean (Standard Deviation); unit: Centimeters (cm)] — This baseline measure describes the length of the participant's laceration (centimeters) at the time of recruitment.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  Centimeters (cm)
    Intention to Treat (ITT): (n = 39, 38, 77) | 2.395 (2.2319) | 2.995 (2.9506) | 2.691 (2.6116)
    Per-Protocol (PP): (n = 35, 36, 71) | 2.389 (2.3241) | 3.056 (3.0184) | 2.727 (2.7003)
Laceration Location: Above Neck [Number; unit: Participants] — This baseline measure describes the number of participants whose laceration was located above the neck i.e., either on the participant's neck or head.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  Participants
    Intention to Treat (ITT) | 25 | 18 | 43
    Per-Protocol (PP) | 22 | 16 | 38
Laceration Location: Below Neck [Number; unit: Participants] — This baseline measure describes the number of participants whose laceration was located above the neck i.e., either on the participant's neck or head.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  Participants
    Intention to Treat (ITT) | 14 | 22 | 36
    Per-Protocol (PP) | 13 | 21 | 34
Weight (kg) [Mean (Standard Deviation); unit: Kilograms (kg)] — This baseline measure describes weight of the participants in kilograms.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  Kilograms (kg)
    Intention to Treat (ITT): (n = 39, 40, 79) | 27.63 (10.271) | 27.67 (17.348) | 27.65 (14.208)
    Per-Protocol (PP): (n = 35, 37, 72) | 27.41 (10.315) | 28.02 (18.002) | 27.72 (14.675)
Triage Vitals: Heart Rate [Mean (Standard Deviation); unit: Beats per Minute (bpm)] — This baseline measure describes the heart rate of participants at triage. Heart rate is measured by the number of contractions of the heart per minute (bpm). Note: not all participants had their heart rate measured at triage.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  Beats per Minute (bpm)
    Intention to Treat (ITT): (n = 13, 14, 27) | 96.54 (15.613) | 102.71 (13.088) | 99.74 (14.42)
    Per-Protocol (PP): (n = 13, 13, 26) | 96.54 (15.613) | 102.00 (13.335) | 99.27 (14.496)
Triage Vitals: Blood Pressure (Systolic) [Mean (Standard Deviation); unit: mm Hg] — This baseline measure describes the blood pressure (systolic) at triage measured in millimeters of mercury (mm Hg). Note: not all participants had their blood pressure (systolic) measured at triage.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  mm Hg
    Intention to Treat (ITT): (n = 10, 9, 19) | 110.9 (10.826) | 115.56 (15.915) | 113.11 (13.300)
    Per-Protocol (PP): (n = 10, 9, 19) | 110.9 (10.826) | 115.56 (15.915) | 113.11 (13.300)
Triage Vitals: Blood Pressure (Diastolic) [Mean (Standard Deviation); unit: mm Hg] — This baseline measure describes the blood pressure (diastolic) at triage measured in millimeters of mercury (mm Hg). Note: not all participants had their blood pressure (diastolic) measured at triage.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  mm Hg
    Intention to Treat (ITT): (n = 10, 9, 19) | 66.00 (12.702) | 73.22 (7.759) | 69.42 (11.007)
    Per-Protocol (PP): (n = 10, 9, 19) | 66.00 (12.702) | 73.22 (7.759) | 69.42 (11.007)
Triage Vitals: Oxygen Saturation [Mean (Standard Deviation); unit: Percent (%)] — This baseline measure describes the oxygen saturation at triage measured in percent (%). Note: not all participants had their oxygen saturation measured at triage.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  Percent (%)
    Intention to Treat (ITT): (n = 9, 9, 18) | 99.00 (1.658) | 99.22 (1.394) | 99.11 (1.491)
    Per-Protocol (PP): (n = 9, 8, 17) | 99.00 (1.658) | 99.13 (1.458) | 99.06 (1.519)
Nasal Congestion [Number; unit: Participants] — This baseline characteristic is a measure of the number of participants who experienced nasal congestion at the time of recruitment.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  Participants
    Intention to Treat (ITT) | 5 | 9 | 14
    Per-Protocol (PP) | 4 | 9 | 13
LET: Lidocaine, Epinephrine and Tetracaine Gel Use [Number; unit: participants] — LET is a combination of lidocaine (4 percent), epinephrine (0.1 percent), and tetracaine (0.5 percent) available for use as a topical anesthetic. This baseline variable describes participants who had LET applied to their wounds prior to sutures.
  This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
  This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
  participants
    Intention to Treat (ITT) | 24 | 26 | 50
    Per-Protocol (PP) | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Intention to Treat (ITT): Modified Yale Preoperative Anxiety Score (mYPAS)
Description: Measurement of patient anxiety used to test effect of anxiolytic pre-medication.The mYPAS consists of 5 items (activity, vocalizations, emotional expressivity, state of apparent arousal, and use of parents). Each item has Likert scale whereby participant's behavior is rated from 1 to 4 (Note: Vocalizations is the only item rated from 1 to 6), with higher numbers indicating the highest severity within that item. Each participant was given a mYPAS score for the "suturing" by two independent raters. These raters watched a digital recording of the participant undergoing suturing and from this digital recording used the mYPAS scale to assign a measurement of the participant's anxiety.
  The mYPAS scale is rated as follows: Final scores = (Activity/4 + Vocal/6 + Emotional/4 + Arousal/4 + Parents/4) X 20. Scores range from 23 to 100 where a lower score is indicative of a lower level of anxiety and a higher is indicative of a higher level of anxiety.
Time Frame: Day 1: During suturing
Population: This is for the Intention to Treat analysis and thus, includes all participants that received the study intervention i.e., intranasal saline or intranasal midazolam.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 34 | 39
units on a scale | 59.9201 (30.2724) | 46.2871 (20.5941)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.026, t-test, 2 sided

2. Primary Outcome: Per-Protocol: Modified Yale Preoperative Anxiety Score (mYPAS)
Description: as for outcome 1
Time Frame: Day 1: During suturing
Population: This is for the per-protocol analysis and thus, includes all participants who fulfill the protocol in the terms of eligibility, all interventions, and outcome assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 35 | 37
units on a scale | 58.7056 (29.8887) | 45.4633 (21.20793)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.036, t-test, 2 sided

3. Secondary Outcome: Intention to Treat (ITT): Modified Yale Preoperative Anxiety Score (mYPAS)
Description: as for outcome 1
Time Frame: Day 1: During Baseline, Intervention & Lidocaine
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 39 | 40
units on a scale
  Baseline (n = 35, 38) | 29.9257 (8.5783) | 32.9461 (9.137)
  Intervention (n = 32, 38) | 45.1373 (20.9071) | 58.5803 (25.6165)
  Lidocaine (n = 34, 36) | 68.8275 (26.1481) | 61.1871 (22.9957)
  Suturing Minus Baseline (n = 33, 38)) | 30.3485 (31.0004) | 13.2166 (18.719)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.151, t-test, 2 sided — This is in reference to the baseline measure
Statistical Analysis 2: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.020, t-test, 2 sided — This is in reference to the intervention measure
Statistical Analysis 3: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.198, t-test, 2 sided — This is in reference to the lidocaine measure
Statistical Analysis 4: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — This is in reference to the difference between the suturing and baseline measures

4. Secondary Outcome: Per-Protocol: Modified Yale Preoperative Anxiety Score (mYPAS)
Description: as for outcome 1
Time Frame: Day 1: Baseline, Intervention & Lidocaine
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 35 | 37
units on a scale
  Baseline (n = 33, 36) | 30.0318 (8.8073) | 32.9736 (9.3917)
  Intervention (n = 30, 36) | 43.0638 (19.5711) | 57.9917 (25.7323)
  Lidocaine (n = 34, 35) | 68.8275 (26.1481) | 60.9596 (23.29024)
  Suturing Minus Baseline (n = 32, 36) | 29.1328 (30.6868) | 12.4897 (18.95566)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.185, t-test, 2 sided — This is in reference to the baseline measure
Statistical Analysis 2: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.011, t-test, 2 sided — This is in reference to the intervention measure
Statistical Analysis 3: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.191, t-test, 2 sided — This is in reference to the lidocaine measure
Statistical Analysis 4: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.008, t-test, 2 sided — This is in reference to the difference between the suturing and baseline measures

5. Secondary Outcome: Intention to Treat (ITT): State Trait Anxiety Inventory (STAI)
Description: Validated measurement of anxiety, to be used to test parental/guardian anxiety at two time points. These time points are before intervention and immediately after suturing (prior to patient discharge from the ER, i.e. same day). The STAI contains 10 items for assessing trait anxiety and 10 for state anxiety. All items are rated on a standard scale ("Not at all", "Somewhat", "Moderately so", "Very much so") with a range of 20 to 80 where higher scores indicate greater anxiety and lower scores indicate lower levels of anxiety.
Time Frame: Day 1: Before intervention and immediately after suturing (prior to patient discharge from the ER, i.e. same day)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 39 | 40
units on a scale
  STAI Pre (n = 36, 37) | 39.3333 (11.1867) | 43.1351 (14.6461)
  STAI Post (n = 37, 40) | 38.3784 (12.7788) | 34.5500 (11.2682)
  STAI Post Minus Pre (n = 35, 37) | -0.5143 (8.8993) | -8.2162 (12.4992)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.004, t-test, 2 sided — This p value is a t-test of the Post STAI minus Pre STAI variable

6. Secondary Outcome: Per-Protocol: State Trait Anxiety Inventory (STAI)
Description: as for outcome 5
Time Frame: Before intervention and immediately after suturing (prior to patient discharge from the ER, i.e. same day)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 35 | 37
units on a scale
  STAI Pre (n = 32, 34) | 39.3438 (11.21522) | 41.7353 (14.2261)
  STAI Post (n = 34, 37) | 38.4118 (12.8184) | 33.7568 (11.2926)
  STAI Post Minus Pre (n = 32, 34) | -0.8750 (9.1643) | -7.6471 (12.4897)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.015, t-test, 2 sided — This p value is in reference to the t-test performed for STAI Post Minus STAI Pre

7. Secondary Outcome: Intention to Treat (ITT): Dartmouth Operative Conditions Scale
Description: A tool to measure the effectiveness and safety of pediatric sedation, regardless of technique used for decreasing anxiety or pain during a procedure. The scale asks the physician to rate patient states (pain/stress, movement, consciousness & sedation side effects) based on observed behaviors (each observed behavior is given a score). The scores are then added together to give a score where -3 to 5 where the lower number is indicative of less anxiety/pain.
Time Frame: Day 1: Immediately after suturing (prior to patient discharge from the ER, i.e. same day)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 37 | 40
units on a scale | 1.92 (1.949) | 1.15 (1.847)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.080, t-test, 2 sided

8. Secondary Outcome: Per-Protocol: Dartmouth Operative Conditions Scale
Description: as for outcome 7
Time Frame: Day 1: Immediately after suturing (prior to patient discharge from the ER, i.e. same day)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 34 | 37
units on a scale | 1.88 (1.966) | 1.08 (1.906)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p = 0.086, t-test, 2 sided

9. Secondary Outcome: Intention to Treat (ITT): Faces Pain Scale-Revised/ FLACC Scale
Description: Faces Pain Scale: Validated self-report tool of pain for participants less than 5 years old. It is a scale that allows one to score the sensation of pain from zero to ten. The scale shows a visuals (faces) for each levels 0, 2, 4, 6, 8 and 10 of the scale. For example, 0 is represented by a "face" visual that expresses no hurt.
  FLACC Scale: Tool to assess pain in children unable to use Faces Pain Scale-revised. The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 (0 represents no pain).
Time Frame: Day 1: immediately after intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 38 | 40
units on a scale | 2.61 (2.605) | 5.25 (2.898)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

10. Secondary Outcome: Per-Protocol: Faces Pain Scale-Revised/ FLACC Scale
Description: as for outcome 9
Time Frame: Day 1: immediately after intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 34 | 37
units on a scale | 2.47 (2.608) | 5.19 (2.895)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Midazolam; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

11. Other Pre Specified Outcome: Time That the Participant Remained in Hospital After Procedure (Mins)
Description: Length of stay in the emergency department, measured from the end of the procedure to the time of discharge.
Time Frame: Day 1: at discharge from emergency department (i.e. same day)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 39 | 40
minutes
  Intentiont to Treat (ITT): (n = 36, 39) | 10.89 (12.673) | 25.41 (26.441)
  Per-Protocol (PP): (n = 33, 37) | 11.24 (13.079) | 25.08 (26.990)

12. Other Pre Specified Outcome: Length of Procedure (Mins)
Description: This is a measure of the length of the procedure (suturing) in minutes.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 39 | 40
minutes
  Intention to Treat (ITT): (n = 36, 39) | 14.72 (7.509) | 23.18 (23.374)
  Per-Protocol (PP): (n = 33, 37) | 15.00 (7.734) | 23.19 (24.014)

13. Other Pre Specified Outcome: Physician's Prediction is Respect to Intervention Drug
Description: This is a measure how how many times the physician was correct in predicting whether the patient received intranasal saline or intranasal midazolam as the intervention drug.
Time Frame: Day 1: physician asked immediately after procedure finished
Measure: Number; unit: Times correct
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 39 | 40
Times correct
  Intention to Treat (ITT): (Total n = 37, 36) | 30 | 31
  Per-Protocol (PP): (Total n = 34, 33) | 28 | 28

14. Other Pre Specified Outcome: Guardian/Parent's Prediction is Respect to Intervention Drug
Description: This is a measure how how many times the parent/guardian was correct in predicting whether the patient received intranasal saline or intranasal midazolam as the intervention drug.
Time Frame: Day 1: parent asked immediately after procedure complete
Measure: Number; unit: Times correct
Arm/Group | Intranasal Saline | Intranasal Midazolam
Number analyzed (Participants) | 39 | 40
Times correct
  Intention to Treat (ITT): (Total n = 35, 38) | 25 | 31
  Per-Protocol (PP): (Total n = 32, 35) | 22 | 28

ADVERSE EVENTS:
Arm/Group | Intranasal Saline | Intranasal Midazolam
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 2/39 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Saline (N=39) | Intranasal Midazolam (N=40)
oxygen saturation less than 92% (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — Not requiring intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes